CLINICAL TRIAL: NCT06073249
Title: Comparison of the Efficacy of Different Nerve Stimulation Methods in Individuals With Chronic Consipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E-10840098-772.02-6150
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Constipation
Keywords: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular vagus stimulation: (Experimental): This non-invasive system is activated by the cutaneous distribution of vagus nerve afferents through the external ear (auricle). Somatosensory innervation is provided by the auricular branch. The name of this device is vagustim device, which consists of a TENS device placed in the outer ear; headphones that can be selected to the size of the individual's ear and a TENS device in which stimulation current is given superficially. In our study, we will perform the application non-invasively by stimulating the branch of the vagus nerve in the auricle. The application time will take 20 minutes.
  Interventions: Other: Auricular vagus stimulation
- Tibial Nerve Stimulation (Active Comparator): The nervus tibialis approaches the surface when it approaches the medial malleolus. In this study, transcutaneous electrical nerve stimulation (TENS) electrodes will be placed under the medial malleolus at the point where the nervus tibialis contacts the surface and approximately bilaterally.
  Interventions: Other: Tibial Nerve Stimulation

INTERVENTIONS:
Other: Auricular vagus stimulation — Non-invasive transcutaneous devices stimulate the vagus nerve via the auricular or carotid artery. It is also used to treat various disorders such as epilepsy, pain and headache. This device stimulates the auricular branch of the vagus nerve non-invasively without any procedure. As a result, it has been found that the pain threshold increases and mechanical pain sensitivity decreases.
  Arms: Auricular vagus stimulation:
Other: Tibial Nerve Stimulation — The sacral plexus provides innervation of the perineal muscle. Its branches (lumbar 4-5 and sacral 1-3) merge to form the nervus ischiadicus, which then divides into two branches. The thick branch of the nervus ischiadicus is the nervus tibialis (lumbar 4-5 and sacral 1-3) and the thin branch is the nervus peroneus communis (lumbar 4-5 and sacral 1-2).
  Arms: Tibial Nerve Stimulation

SUMMARY:
Consipation is the most common digestive complaint in the general population. The normal frequency of defecation ranges from a minimum of three times a week to a maximum of two times a day.

DETAILED DESCRIPTION:
Constipation is one of the most common health problems in the geriatric population, negatively affecting the physical and emotional status of individuals. Constipation can be classified into three main groups: normal transit time constipation, slow transit time constipation and dyssynergic defecation disorders .

Treatment in chronic constipation should be directed towards the underlying cause. In the treatment of chronic constipation, lifestyle modifications and physiotherapy are the first, pharmacologic treatment is the second, and surgical treatment is the third. Physiotherapy modalities such as defecation training, classical massage, electrical stimulation, anorectal biofeedback and exercise training can be used in the treatment of chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 ages Female
* Rome III diagnostic criteria

Exclusion Criteria:

* Severe heart or kidney diseaseprevious gastrointestinal, spinal or pelvic surgery other than cholecystectomy, hysterectomy or appendectomy neurological diseases such as multiple sclerosis, stroke, Parkinson's disease or spinal injury,
* Impaired awareness (mini-mental score < 15),
* Legal blindness, pregnancy,
* Rectal prolapse
* Anal fissure and altered constipation and diarrhea pattern.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — woman
Enrollment: 18 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Bristol Stool Scale (BGS) | 4 weeks
  n the scale developed by Lewis and Heaton in 1990, the type of stool is classified in 7 different groups. In the Bristol Stool Scale, the transit time of stool through the intestine is evaluated over seven different stool types. According to BGS, 1-2 points are shown as "hard stool", 3-4-5 points as "normal stool" and 6-7 points as "soft-watery stool
Pelvic Pain Impact Questionnaire | 4 weeks
  The questionnaire for clinical assessment of the impact of pelvic pain on women consists of 10 questions. However, the first 8 questions are scored. The range of scores to be obtained from the questionnaire varies between 1- 32. As the score value to be obtained from the questionnaire increases, the degree of functional limitation of pelvic pain on the person increases.
Constipation Severity Scale | 4 weeks
  Constipation Severity Scale (CSS): The CSS is a scale for determining the frequency, intensity and difficulty/difficulty during defecation. This scale can also be used to measure symptoms of constipation. The scale includes 16 questions.The minimum total score that can be obtained from the KCS is 0 and the maximum score is 73. A high score on the scale indicates that the symptoms are serious. The highest score that can be obtained from the five-point Likert-type scale is 140 and the lowest score is 28. As the scores obtained from the scale increase, it is thought that the quality of life is negatively affected
Superficial Electromyography Biofeedback | 4 weeks
  For the assessment, the display scale was used as visual feedback and the signal sound, which increases or decreases with changing muscle activity, was used as sensory feedback. Before starting the treatment, the desired goal for the patient is determined. 10 seconds of contraction and relaxation is practiced with the "set target" feature on the device and the average target is determined.
Autonomic nervous system device | 4 weeks
  The Polar H10 device is a heart rate sensor with the gold standard in high precision and accuracy that comes with a wearable chest strap. It can connect to multiple training devices via Bluetooth and ANT+. The device comes with a soft, adjustable sensor that contacts the chest to capture heart rate in real time.
  The study will evaluate the autonomic nervous system with the Polar H10 device. The data will be recorded by connecting the device to a smart phone via bluetooth and the software supported by the device will be used to analyze the data. The participant will be in a sitting position and a measurement will be made for 1 minute. In order for the device to make an accurate measurement, the electrode surface must be wetted before each measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No